CLINICAL TRIAL: NCT02416024
Title: Arterial Stiffness as a Predictor of Refractory Hypotension After Induction of General Anesthesia in Patients Chronically Treated With Angiotensin-converting Enzyme Inhibitors
Brief Title: Arterial Stiffness and General Anesthesia Induced Hypotension in Patients on Angiotensin-converting Enzyme Inhibitors
Status: Completed | Type: Observational
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Kenichi Ueda, Clinical Associate Professor, University of Iowa
Other Study IDs: 201308815
Record Dates: First submitted 2015-04-06; First posted 2015-04-14 (Estimated); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Hypotension; Arterial Stiffness
Keywords: angiotensin converting enzyme inhibitor; anesthesia
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- No Refractory hypotension group: Patient who did not require more than 200 mcg of phenylephrine to maintain systemic blood pressure during 10 minutes after induction of general anesthesia.
  Interventions: Device: SphygmoCor system
- Control: Patient who required more than 200 mcg of phenylephrine to maintain systemic blood pressure during 10 minutes after induction of general anesthesia
  Interventions: Device: SphygmoCor system

INTERVENTIONS:
Device: SphygmoCor system — Carotid-femoral pulse wave velocity (cfPWV) will be determined by applanation tonometry using the Sphygmocor system by sequentially recording ECG-gated carotid and femoral artery waveforms. Pulse wave signals will be recorded by tonometers positioned at the base of the right common carotid artery and over the right femoral artery. The time (t) between the feet of simultaneously recorded waves will be determined as the mean of 10 consecutive cardiac cycles. PWV is calculated by the system software from the distance between measurement points (D) and the measured time delay (t) as follows: cfPWV = D/Δt (m/s) where D is distance in meters and t is the time interval in seconds.

SUMMARY:
Induction of general anesthesia to the patient could be a challenging period of anesthesia management. Due to autonomic system suppression, hemodynamic fluctuation, such as hypotension or hypertension, is commonly seen during this period. Furthermore, it has been observed that a fraction of patients who develop hypotension may be refractory to vasoactive medications to attempt to restore the systemic arterial blood pressure back to an acceptable level.

Previous studies have shown that patients chronically taking angiotensin converting enzyme (ACE) inhibitors have a higher incidence of developing hypotension under general anesthesia as well as being refractory to adrenergic vasoconstrictor medications given to help restore systemic blood pressure. Interestingly, not all patients taking ACE inhibitors have shown the described hemodynamic response after induction of general anesthesia. Therefore, investigators are attempting to identify what changes in vascular physiology in those patients may contribute to acute refractory systemic hypotension. Specifically, investigators wish to explore whether differences in baseline levels of arterial stiffness potentially contribute to this phenomenon. Arterial applanation tonometry is a non-invasive technique that has been shown to reliably provide indices of arterial stiffness. In the proposed project, applanation tonometry will be performed on the right carotid and femoral arteries to assess carotid-femoral pulse wave velocity, a surrogate for aortic stiffness. (SphygmoCor system, AtCor Medical, Sydney, Australia) The measurement will be obtained before induction of general anesthesia in the pre-surgical area. During induction of general anesthesia with standard induction agents, brachial blood pressure will be measured by a cuff every minute up to 10 minutes after tracheal intubation. A hypotensive response to anesthesia will be defined by a systolic arterial blood pressure below 90mmHg upon induction. Hypotensive patients that do not respond to vasoconstrictor medications (i.e. requires more than 200 mcg phenylephrine to maintain systolic arterial blood pressure above 90 mmHg) will be classified as 'refractory hypotensive." Using non-invasive applanation tonometry, we will be able to examine if aortic stiffness has a propensity to become refractory hypotension after induction of general anesthesia. This information will potentially help identify future patients that might be at greater risk of developing refractory hypotension in response to induction of general anesthesia.

DETAILED DESCRIPTION:
Background: Induction of anesthesia consists with administration of anesthetics followed by endotracheal intubation. During the induction of anesthesia moderate hemodynamic disturbances (either systemic arterial hyper- or hypo-tension) are common due to concurrent autonomic nervous system suppression and from the stress response from endotracheal intubation. Previous studies demonstrate that patients chronically treated with angiotensin converting enzyme (ACE)-inhibitors have higher incidence of developing hypotension after induction of general anesthesia, which typically, can be restored with small doses of adrenergic drugs such as phenylephrine (100 to 200 mcg) to acceptable blood pressure levels. However, some patients that develop hypotension may be refractory to those medications, which in turn poses a significant challenge in controlling the hemodynamics of patients. The consequence of the severe hypotension could be canceled surgery, ischemic stroke, myocardial infarction or even death.

Interestingly, this refractory systemic hypotension does not occur in all anesthetized patients prescribed ACE inhibitors. Notably, easily treatable systemic arterial hypotension after induction of general anesthesia is not a clinical problem. Critical issue arises only if the patient under general anesthesia does not respond to therapeutic doses of adrenergic agonists. Therefore, identifying patients who will demonstrate refractory hypotension after the induction of general anesthesia is a novel idea and has significant clinical implications for peri-operative blood pressure control by anesthesiologists.

Thus, the overall goals of the proposed research will be to use preoperative non-invasive measures of vascular stiffness to predict which patients might be at risk for severe hypotension that is refractory to adrenergic vasoconstrictor medications following induction of general anesthesia in patients chronically treated with angiotensin-converting enzyme inhibitors.

Method/Design: The study will be human subject non-randomized observational study. This study will be conducted at day of surgery administration area and main operation room at University of Iowa Hospitals and clinics. Arterial stiffness will be measured at day of surgery administration area prior to the surgery.

Carotid-Femoral Pulse Wave Velocity (Aortic Stiffness). Carotid-femoral pulse wave velocity (cfPWV) will be determined by applanation tonometry using the Sphygmocor system by sequentially recording ECG-gated carotid and femoral artery waveforms. Pulse wave signals will be recorded by tonometers positioned at the base of the right common carotid artery and over the right femoral artery. The time (t) between the feet of simultaneously recorded waves will be determined as the mean of 10 consecutive cardiac cycles. PWV is calculated by the system software from the distance between measurement points (D) and the measured time delay (t) as follows: cfPWV = D/Δt (m/s) where D is distance in meters and t is the time interval in seconds.

Prior to induction intravenous fluid administration will be restricted to less than 500 ml. A standardized protocol will be followed which is commonly used by anesthesia providers. Prior to induction of anesthesia, in addition to ASA standard monitors, neuromuscular twitch monitor and Entropy monitor will be attached to the patient. Induction agents will include 1.5mg/kg propofol, 2µg/kg fentanyl, 100mg lidocaine, and 0.6 mg/kg rocuronium of lean body weight. Inhaled anesthetic will be sevoflurane at 0.5 MAC with 5L/min of 100% oxygen starting at mask ventilation till 10 minutes after tracheal intubation. Blood pressure will be measured by a brachial cuff prior to induction and every minute after intubation for 10 minutes. If the systolic pressure drops below 90 mmHg or more than 25% from baseline, the patient will be classified in the study as "Hypotensive." Conversely, if the patient's systolic blood pressure does not drop below 90 mmHg more than 25% from baseline within 10 minutes of intubation, the patient will be classified as "Not Hypotensive." If the patient's systolic blood pressure rises above 25% the baseline value, the anesthesiologist will administer a bolus of 0.5mg/kg of propofol. This bolus will be repeated after the minute blood pressure evaluations until the systolic blood pressure back to the baseline value. These patients will be classified as "Not Hypotensive," but the administration of propofol will be noted. In attempt to bring systolic blood pressure up to above 90 mmHg or more than 25% from baseline in "hypotensive" patients, the anesthetic provider will use 100µg phenylephrine (or 5mg ephedrine if heart rate < 50bpm) within 10 minutes of intubation. If over 200µg phenylephrine (10mg ephedrine) has been used without a return of the systolic brachial blood pressure >90 mmHg or more than 25% from baseline, the patient will be classified in the study as "Refractory Hypotensive." The study environment will be ended and the provider can use whatever vasoactive drugs they deem appropriate, including more phenylephrine, ephedrine, epinephrine, norepinephrine, or vasopressin, and/or fluid bolus. The total given doses of each vasopressor medication will be recorded. Anesthetic induction, blood pressure measurements, and medication to correct low and high blood pressure as described above are all part of the patients' standard clinical procedures as performed by the anesthesiologist. The patients who required more than 2 times laryngoscopy, required other than standard anesthetics, or entropy >70 or <30, will be exclude from data analysis.

ELIGIBILITY:
Inclusion Criteria:

* There will be three study populations. The first study population will include 60 adult patients over 50 years old and on ACE inhibitors for more than 3 months, scheduled for surgery under general anesthesia in the second case in the Main Operating Room at the UIHC. Patients who are taking angiotensin receptor inhibitors will not be enrolled for the study.

The second study population will include 20 adult patients over 50 years old who are not taking an ACE inhibitor and are currently taking a beta blocker, a calcium channel blocker, or a diuretic for more than 3 months, scheduled for surgery under general anesthesia in the Main Operating Room at the UIHC.

Exclusion Criteria:

We will exclude patients with diabetes (on insulin therapy), renal insufficiency (Cr>2.0), history of arterial bypass (i.e. F-F bypass), history of carotid endoarterectomy, angiotensin receptor inhibitor medication, heart rate <40 bpm or >100 bpm, atrial fibrillation/flutter, history of ischemic stroke, transient ischemic attack, myocardial infarction or coronary revascularization (any type) within 6 months, known left main or 3-vessel coronary disease positive myocardial perfusion study without subsequent revascularization, angina or heart failure (>3 NYHA) class 3, known left ventricle ejection fraction <30%, pulmonary hypertension (PA systolic >50mmHg), right ventricle dysfunction, or a preoperative systolic blood pressure of >180 mmHg or <110 mmHg within 1 month prior to surgery.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who are going under surgery with age between 50 - 85
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2013-08; Primary Completion 2018-06 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Comparison of Vascular Stiffness between refractory hypotension and non-refractory hypotension group | within one hour
  The study is aimed to compare arterial stiffness between patients develop refractory hypotension and do not develop refractory hypotension after administration of anesthetics in preparation for surgery of patients older than 60 years of age and with a prescription/current use of ACE-inhibitors. Arterial stiffness will be measured by pulse wave velocity (m/s) with a SphygmoCor® device (Atcor, Sydney, Australia)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

REFERENCES:
- [Result] Gasecki D, Rojek A, Kwarciany M, Kowalczyk K, Boutouyrie P, Nyka W, Laurent S, Narkiewicz K. Pulse wave velocity is associated with early clinical outcome after ischemic stroke. Atherosclerosis. 2012 Dec;225(2):348-52. doi: 10.1016/j.atherosclerosis.2012.09.024. Epub 2012 Oct 3. PMID 23083680
- [Result] Mitchell GF, Hwang SJ, Vasan RS, Larson MG, Pencina MJ, Hamburg NM, Vita JA, Levy D, Benjamin EJ. Arterial stiffness and cardiovascular events: the Framingham Heart Study. Circulation. 2010 Feb 2;121(4):505-11. doi: 10.1161/CIRCULATIONAHA.109.886655. Epub 2010 Jan 18. PMID 20083680
- [Result] Blann AD, Kuzniatsova N, Lip GY. Inflammation does not influence arterial stiffness and pulse-wave velocity in patients with coronary artery disease. J Hum Hypertens. 2013 Oct;27(10):629-34. doi: 10.1038/jhh.2013.17. Epub 2013 Mar 28. PMID 23535991
- [Result] Ozturk S, Baltaci D, Ayhan SS, Durmus I, Gedikli O, Soyturk M, Yazici M, Celik S. Assessment of the relationship between aortic pulse wave velocity and aortic arch calcification. Turk Kardiyol Dern Ars. 2012 Dec;40(8):683-9. doi: 10.5543/tkda.2012.83707. PMID 23518881
- [Result] Dangardt F, Chen Y, Berggren K, Osika W, Friberg P. Increased rate of arterial stiffening with obesity in adolescents: a five-year follow-up study. PLoS One. 2013;8(2):e57454. doi: 10.1371/journal.pone.0057454. Epub 2013 Feb 22. PMID 23451232
- [Result] Nordstrand N, Gjevestad E, Hertel JK, Johnson LK, Saltvedt E, Roislien J, Hjelmesaeth J. Arterial stiffness, lifestyle intervention and a low-calorie diet in morbidly obese patients-a nonrandomized clinical trial. Obesity (Silver Spring). 2013 Apr;21(4):690-7. doi: 10.1002/oby.20099. PMID 23712971
- [Result] Alecu C, Cuignet-Royer E, Mertes PM, Salvi P, Vespignani H, Lambert M, Bouaziz H, Benetos A. Pre-existing arterial stiffness can predict hypotension during induction of anaesthesia in the elderly. Br J Anaesth. 2010 Nov;105(5):583-8. doi: 10.1093/bja/aeq231. Epub 2010 Aug 26. PMID 20798172